CLINICAL TRIAL: NCT01380262
Title: Prospective Phase II Study on Skin Toxicity on Low-Dose Doxycycline in Metastatic Colorectal Cancer Patients During Cetuximab and Panitumumab Treatment
Brief Title: Pre-emptive Low-dose Doxycycline During Anti-EGFR Treatment
Acronym: STLDD-1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Maria Sklodowska-Curie National Research Institute of Oncology (Other)
Responsible Party: Maria Sklodowska-Curie Memorial Cancer Center, Institute of Oncology, Maria Sklodowska-Curie Memorial Cancer Center, Institute of Oncology
Other Study IDs: STLDD-1
Record Dates: First submitted 2011-06-22; First posted 2011-06-27 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Colorectal Cancer; Skin Toxicities
Keywords: Colorectal Cancer; Skin Rash; Pre-emptive treatment; Doxycycline; Anti-EGFR antibody; Cetuximab; Panitumumab
MeSH Terms: conditions — Colorectal Neoplasms; Exanthema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Low Dose Doxycycline: Patients with metastatic colorectal cancer, qualified to either cetuximab or panitumumab based systemic treatment (either monotherapy or with chemotherapy) receiving a 100 mg of doxycycline daily

SUMMARY:
Up to 60% of patients with metastatic colorectal cancer can be treated with one of monoclonal antibodies targeted against epidermal growth factor receptor (EGFR). This treatment is associated with a specific spectrum of toxicity: acne-like rash from limited up to erythema, often with severe pruritus, sometimes combined with other types of skin toxicities (hair and nail changes). Previously in STEPP study investigators shown that pre-emptive treatment with oral doxycycline (200 mg daily), topical steroids and sun blockers reduces the number of more severe skin side effects of panitumumab.

The study is designed to described the profile of skin toxicity of EGFR blocking drugs combined with low-dose doxycycline (100 mg daily) used in the pre-emptive manner.

DETAILED DESCRIPTION:
Patients with metastatic colorectal cancer treated with cetuximab or panitumumab usually develop the skin toxicity which can impair patients' quality of life as well as limit the treatment. We designed this trial to assess the effect of simplified protocol of pre-emptive treatment on the observed skin toxicities during cetuximab and panitumumab treatment of colorectal cancer.

The study is a cohort observational, single center study which should result in estimation of particular types of toxicities, especially occurence of more severe (grade 2 and 3) side effects and assess the tolerance of doxycyline in the prolonged administration.

The observation in the study is biweekly and is continued up to 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of metastatic colorectal cancer,
* previously qualified to either cetuximab or panitumumab,
* written consent.

Exclusion Criteria:

* previous administration of cetuximab or panitumumab,
* contradictions to receive oral doxycycline.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic colorectal cancer, qualified to either cetuximab or panitumumab based systemic treatment (either monotherapy or with chemotherapy) receiving a 100 mg of doxycycline daily.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2010-06; Primary Completion 2011-09 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
number of patients with a severe skin toxicity | 8 weeks

SECONDARY OUTCOMES:
total occurence of skin toxicities | 8 weeks
  analyzed for weeks: 2, 4, 6 and 8 separetly
number of patients with delayed administration of cetuximab or panitumumab due to severe skin toxicity | 8 weeks
quality of life assessed with DLQI | 8 weeks
  assessed as a correlation to severeness of skin toxicities

CONTACTS AND LOCATIONS:
Overall Officials: Lucjan S Wyrwicz, MD,PhD, Principal Investigator — Maria Sklodowska-Curie National Research Institute of Oncology
Locations (1):
- Department of Gastrointestinal Cancer, Maria Sklodowska-Curie Memorial Cancer Center, Institute of Oncology, Warsaw, Masovian Voivodeship, Poland